CLINICAL TRIAL: NCT00882999
Title: Multiple Subcutaneous Doses of LY2127399, an Anti-BAFF Human Antibody, in Subjects With Relapsing-Remitting Multiple Sclerosis
Brief Title: A Study of Participants With Relapsing-Remitting Multiple Sclerosis (RRMS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12778; H9B-MC-BCDJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Relapsing; Remitting; Multiple Sclerosis; Multiple; Sclerosis; MS; LY2127399
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Recurrence; Multiple Sclerosis; Sclerosis | interventions — tabalumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Placebo (Placebo Comparator): Injection: Every 4 weeks in the placebo arm for 24 weeks (Weeks 0, 4, 8, 12, 16, and 20) for a total of 6 doses. Every 4 weeks in the LY2127399 arms [4 milligrams (mg) LY2127399 / 12 weeks and 120 mg LY2127399 / 12 weeks] for 24 weeks (except Week 0 and Week 12).
  Interventions: Drug: Placebo
- 4 mg LY2127399 / 4 weeks (Experimental): Injection: 6 doses, one every 4 weeks for 24 weeks.
  Interventions: Drug: LY2127399
- 40 mg LY2127399 / 4 weeks (Experimental): Injection: 6 doses, one every 4 weeks for 24 weeks.
  Interventions: Drug: LY2127399
- 120 mg LY2127399 / 4 weeks (Experimental): Injection: 6 doses, one every 4 weeks for 24 weeks.
  Interventions: Drug: LY2127399
- 4 mg LY2127399 / 12 weeks (Experimental): Drug: LY2127399 Injection: 2 doses, one every 12 weeks for 24 weeks.
  Drug: Placebo Injection: Every 4 weeks for 24 weeks (except Week 0 and Week 12).
  Interventions: Drug: LY2127399; Drug: Placebo
- 120 mg LY2127399 / 12 weeks (Experimental): Drug: LY2127399 Injection: 2 doses, one every 12 weeks for 24 weeks.
  Drug: Placebo Injection: Every 4 weeks for 24 weeks (except Week 0 and Week 12).
  Interventions: Drug: LY2127399; Drug: Placebo
- 12 mg LY2127399 / 4 weeks (Experimental): Injection: 6 doses, one every 4 weeks for 24 weeks.
  Interventions: Drug: LY2127399

INTERVENTIONS:
Drug: LY2127399 — Administered via Injection
  Arms: 12 mg LY2127399 / 4 weeks; 120 mg LY2127399 / 12 weeks; 120 mg LY2127399 / 4 weeks; 4 mg LY2127399 / 12 weeks; 4 mg LY2127399 / 4 weeks; 40 mg LY2127399 / 4 weeks
Drug: Placebo — Administered via Injection
  Arms: 120 mg LY2127399 / 12 weeks; 4 mg LY2127399 / 12 weeks; Placebo

SUMMARY:
To look at the ability of LY2127399 to reduce magnetic resonance imaging (MRI) lesions at 12, 16, 20, and 24 weeks compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* 18 through 64 years of age diagnosed with RRMS, who can walk without aid or rest for at least 200 meters (approximately 1/10 of a mile).
* Women who can become pregnant must use birth control.

Exclusion Criteria:

* Have had a live vaccination within 12 weeks before randomization, or intend to have a live vaccination during the course of the study.
* Have had had recent surgery or are scheduled to have surgery during the study.
* Are immunocompromised or have evidence of active infection [such as hepatitis, tuberculosis or, human immunodeficiency virus (HIV)].
* Have been on certain drugs that are being studied for RRMS or have recently received prescription drugs to treat RRMS.
* Have had a recent serious infection.
* Have serious or uncontrolled illnesses other than RRMS.
* Have clinically significant blood test values.
* Have multiple or severe drug allergies.
* Have contraindications for MRI "scanning" or claustrophobia (fear of an enclosed space) that cannot be managed.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 245 (Actual)
Dates: Start 2009-04; Primary Completion 2011-02 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon- Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST, Study Director — Eli Lilly and Company
Locations (63):
- United States (27):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fullerton, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Naples, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plantation, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sarasota, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Northbrook, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kansas City, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Biddeford, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Farmington Hills, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Schenectady, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Akron, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Green, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greensburg, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Franklin, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lubbock, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Round Rock, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newport News, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roanoke, Virginia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sofia, Bulgaria
- Czechia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pardubice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nîmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
- Hungary (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Győr
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gyula
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Litwinsky, Israel
- Poland (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gliwice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grodzisk Mazowiecki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow-Nowa Huta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş, Romania
- Russia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kazan'
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kemerovo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
- Serbia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belgrade
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niš
- Slovakia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bratislava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Košice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spišská Nová Ves
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Žilina
- Ukraine (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dnipro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Donetsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ivano-Frankivsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kharkiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vinnytsia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included 24 weeks of treatment and 24 weeks of follow-up. If necessary, participants had additional long-term follow-up for peripheral blood B cell monitoring (up to Week 108). Participants who completed study treatment (24 weeks) and the initial study follow-up (24 weeks) were considered study completers.
Groups:
- 4 mg LY2127399 Q4W: LY2127399: 4 milligrams (mg) subcutaneous injection once every 4 weeks (Q4W) for 24 weeks (Weeks 0, 4, 8, 12, 16, and 20).
- 12 mg LY2127399 Q4W: LY2127399: 12 mg subcutaneous injection Q4W for 24 weeks.
- 40 mg LY2127399 Q4W: LY2127399: 40 mg subcutaneous injection Q4W for 24 weeks.
- 120 mg LY2127399 Q4W: LY2127399: 120 mg subcutaneous injection Q4W for 24 weeks.
- 4 mg LY2127399 Q12W: LY2127399: 4 mg subcutaneous injection every 12 weeks (Q12W) for 24 weeks (Weeks 0 and 12).
  Placebo: Subcutaneous injection Q4W for 24 weeks except (Weeks 0 and 12).
- 120 mg LY2127399 Q12W: LY2127399: 120 mg subcutaneous injection Q12W for 24 weeks (Weeks 0 and 12).
  Placebo: Subcutaneous injection Q4W for 24 weeks except (Weeks 0 and 12).
- Placebo: Placebo: Subcutaneous injection Q4W for 24 weeks.
Period: Overall Study
Arm/Group | 4 mg LY2127399 Q4W | 12 mg LY2127399 Q4W | 40 mg LY2127399 Q4W | 120 mg LY2127399 Q4W | 4 mg LY2127399 Q12W | 120 mg LY2127399 Q12W | Placebo
Started | 35 | 34 | 34 | 36 | 36 | 35 | 35
Received Any Amount of Study Drug | 35 | 34 | 34 | 36 | 36 | 35 | 35
Completed Study Treatment | 29 | 29 | 31 | 33 | 29 | 30 | 31
Completed | 27 | 26 | 30 | 31 | 28 | 28 | 27
Not Completed | 8 | 8 | 4 | 5 | 8 | 7 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 6 | 3 | 3 | 6 | 5 | 5
Not completed — Lost to Follow-up | 0 | 1 | 1 | 2 | 1 | 1 | 2
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 4 mg LY2127399 Q4W: LY2127399: 4 mg subcutaneous injection Q4W for 24 weeks (Weeks 0, 4, 8, 12, 16, and 20).
- 4 mg LY2127399 Q12W: LY2127399: 4 mg subcutaneous injection Q12W for 24 weeks (Weeks 0 and 12).
  Placebo: Subcutaneous injection Q4W for 24 weeks (except Weeks 0 and 12).
- 120 mg LY2127399 Q12W: LY2127399: 120 mg subcutaneous injection Q12W for 24 weeks (Weeks 0 and 12).
  Placebo: Subcutaneous injection Q4W for 24 weeks (except Weeks 0 and 12).
- Total: Total of all reporting groups
Arm/Group | 4 mg LY2127399 Q4W | 12 mg LY2127399 Q4W | 40 mg LY2127399 Q4W | 120 mg LY2127399 Q4W | 4 mg LY2127399 Q12W | 120 mg LY2127399 Q12W | Placebo | Total
Number analyzed (Participants) | 35 | 34 | 34 | 36 | 36 | 35 | 35 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (10.23) | 43.1 (10.06) | 40.8 (10.78) | 40.8 (11.10) | 43.1 (10.62) | 39.0 (10.16) | 40.3 (12.02) | 41.3 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 27 | 21 | 27 | 24 | 24 | 169
  Male | 11 | 12 | 7 | 15 | 9 | 11 | 11 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 4
  Not Hispanic or Latino | 35 | 34 | 34 | 35 | 34 | 35 | 34 | 241
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 0 | 0 | 2 | 6 | 2 | 3 | 17
  White | 31 | 34 | 34 | 34 | 30 | 33 | 32 | 228
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 10 | 15 | 15 | 22 | 18 | 14 | 108
  Slovakia | 5 | 5 | 3 | 6 | 3 | 4 | 6 | 32
  Ukraine | 2 | 2 | 1 | 1 | 0 | 2 | 0 | 8
  Israel | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Russia | 2 | 1 | 4 | 3 | 1 | 1 | 1 | 13
  France | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 4
  Czechia | 0 | 2 | 1 | 0 | 0 | 2 | 1 | 6
  Hungary | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 5
  Poland | 3 | 5 | 2 | 3 | 5 | 2 | 3 | 23
  Romania | 1 | 1 | 1 | 2 | 0 | 1 | 2 | 8
  Bulgaria | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3
  Finland | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 5
  Germany | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Canada | 4 | 2 | 5 | 3 | 4 | 3 | 4 | 25
Time Since Onset Of First Symptoms [Mean (Standard Deviation); unit: years] | 8.5 (7.81) | 9.4 (6.96) | 9.2 (7.49) | 8.9 (9.52) | 7.8 (5.93) | 9.2 (8.48) | 7.4 (6.70) | 8.6 (7.58)
Time Since First Diagnosis [Mean (Standard Deviation); unit: years] | 5.9 (7.19) | 6.3 (6.19) | 5.4 (6.67) | 5.0 (7.50) | 5.0 (5.03) | 6.0 (5.73) | 3.8 (4.88) | 5.3 (6.21)
Number Of Relapses In Past Year [Mean (Standard Deviation); unit: relapses] | 1.4 (1.26) | 1.3 (0.51) | 1.4 (0.73) | 1.2 (0.56) | 1.4 (1.11) | 1.5 (0.89) | 1.5 (1.38) | 1.4 (0.97)
Number of Gadolinium (Gd)-Enhancing T1-Weighted Lesions [Mean (Standard Deviation); unit: lesions] — Lesions were measured through Gd-enhancing T1-weighted magnetic resonance imaging (MRI) scans.
  lesions | 1.1 (2.64) | 0.5 (0.93) | 1.1 (1.91) | 1.4 (2.60) | 1.3 (2.41) | 1.2 (2.11) | 1.2 (2.08) | 1.1 (2.16)
Volume of T2-Weighted Lesions [Mean (Standard Deviation); unit: milliliters (mL)] — Lesions were measured through T2-weighted proton density MRI scans.
  milliliters (mL) | 8.5 (10.53) | 7.8 (9.21) | 6.6 (7.92) | 9.0 (11.90) | 10.1 (13.90) | 7.1 (7.66) | 7.0 (8.07) | 8.0 (10.10)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Gd-Enhancing T1-Weighted MRI Lesions Per Scan Averaged During Weeks 12, 16, 20, and 24
Description: Lesions were measured using Gd-enhancing T1-weighted MRI scans. The number of T1-weighted lesions per scan was obtained from the number of T1-weighted lesions observed during a specified week divided by the number of scans performed that same week. To obtain the number of T1-weighted lesions per scan averaged during Weeks 12, 16, 20, and 24, the number of lesions per scan at each week was summed and then divided by the number of visits with non-missing lesion counts.
Time Frame: Weeks 12, 16, 20, and 24
Population: Randomized participants who had a Gd-enhancing T1-weighted MRI lesion for at least 1 time point among Weeks 12, 16, 20, or 24.
Measure: Mean (Standard Deviation); unit: lesions per scan
Arm/Group | 4 mg LY2127399 Q4W | 12 mg LY2127399 Q4W | 40 mg LY2127399 Q4W | 120 mg LY2127399 Q4W | 4 mg LY2127399 Q12W | 120 mg LY2127399 Q12W | Placebo
Number analyzed (Participants) | 34 | 31 | 31 | 36 | 36 | 34 | 33
lesions per scan | 1.819 (3.312) | 0.710 (1.103) | 1.237 (1.999) | 1.477 (2.834) | 2.319 (4.145) | 1.422 (3.058) | 1.758 (3.615)

2. Secondary Outcome: Change From Baseline in Number of Gd-Enhancing T1-Weighted MRI Lesions Per Scan
Description: Lesions were measured using Gd-enhancing T1-weighted MRI scans. The number of T1-weighted lesions per scan was obtained from the number of T1-weighted lesions observed during a specified week divided by the number of scans performed that same week. Least squares (LS) mean was calculated using an analysis of variance (ANOVA).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 36, and 48
Population: Randomized participants who had a Gd-enhancing T1-weighted MRI assessment at the specified time points.
Measure: Least Squares Mean (Standard Error); unit: lesions per scan
Arm/Group | 4 mg LY2127399 Q4W | 12 mg LY2127399 Q4W | 40 mg LY2127399 Q4W | 120 mg LY2127399 Q4W | 4 mg LY2127399 Q12W | 120 mg LY2127399 Q12W | Placebo
Number analyzed (Participants) | 34 | 33 | 31 | 36 | 36 | 34 | 34
lesions per scan
  Week 4: number analyzed (Participants) | 34 | 31 | 31 | 36 | 35 | 34 | 34
  Week 4 | -0.2 (0.09) | -0.3 (0.09) | -0.3 (0.09) | -0.3 (0.09) | 0.0 (0.09) | -0.3 (0.09) | -0.1 (0.09)
  Week 8: number analyzed (Participants) | 33 | 33 | 31 | 35 | 36 | 32 | 34
  Week 8 | -0.2 (0.10) | -0.3 (0.10) | -0.3 (0.10) | -0.3 (0.09) | -0.0 (0.09) | -0.2 (0.10) | -0.2 (0.09)
  Week 12: number analyzed (Participants) | 32 | 28 | 30 | 35 | 36 | 31 | 32
  Week 12 | -0.1 (0.10) | -0.3 (0.11) | -0.1 (0.10) | -0.2 (0.10) | -0.1 (0.10) | -0.1 (0.10) | -0.2 (0.10)
  Week 16: number analyzed (Participants) | 33 | 27 | 30 | 34 | 31 | 31 | 31
  Week 16 | -0.2 (0.10) | -0.3 (0.11) | -0.2 (0.10) | -0.2 (0.09) | -0.0 (0.10) | -0.2 (0.10) | -0.2 (0.10)
  Week 20: number analyzed (Participants) | 27 | 28 | 30 | 34 | 30 | 32 | 32
  Week 20 | -0.3 (0.10) | -0.4 (0.10) | -0.2 (0.10) | -0.1 (0.09) | -0.1 (0.10) | -0.3 (0.09) | -0.2 (0.09)
  Week 24: number analyzed (Participants) | 28 | 28 | 29 | 32 | 28 | 30 | 31
  Week 24 | -0.2 (0.10) | -0.4 (0.10) | -0.2 (0.10) | -0.3 (0.09) | -0.3 (0.10) | -0.3 (0.09) | -0.2 (0.09)
  Week 36: number analyzed (Participants) | 26 | 26 | 31 | 32 | 28 | 31 | 29
  Week 36 | -0.3 (0.10) | -0.4 (0.10) | -0.3 (0.09) | -0.2 (0.09) | -0.2 (0.10) | -0.2 (0.09) | -0.2 (0.10)
  Week 48: number analyzed (Participants) | 26 | 25 | 27 | 31 | 26 | 25 | 24
  Week 48 | -0.4 (0.09) | -0.5 (0.09) | -0.4 (0.09) | -0.3 (0.08) | -0.4 (0.09) | -0.3 (0.09) | -0.3 (0.10)

3. Secondary Outcome: Total Number of New Gd-Enhancing T1-Weighted MRI Lesions Per Scan
Description: Lesions were measured using Gd-enhancing T1-weighted MRI scans. The number of new T1-weighted lesions per scan was obtained from the number new T1-weighted lesions observed during a specified week divided by the number of scans performed that same week.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 36, and 48
Population: Randomized participants who had a Gd-enhancing T1-weighted MRI assessment at the specified time points.
Measure: Mean (Standard Deviation); unit: lesions per scan
Arm/Group | 4 mg LY2127399 Q4W | 12 mg LY2127399 Q4W | 40 mg LY2127399 Q4W | 120 mg LY2127399 Q4W | 4 mg LY2127399 Q12W | 120 mg LY2127399 Q12W | Placebo
Number analyzed (Participants) | 34 | 33 | 31 | 36 | 36 | 34 | 34
lesions per scan
  Week 4: number analyzed (Participants) | 34 | 31 | 31 | 36 | 35 | 34 | 34
  Week 4 | 1.1 (1.67) | 0.6 (1.09) | 0.6 (1.23) | 0.5 (1.11) | 1.9 (3.00) | 0.9 (1.71) | 1.4 (2.44)
  Week 8: number analyzed (Participants) | 33 | 33 | 31 | 35 | 36 | 32 | 34
  Week 8 | 1.4 (2.52) | 0.6 (1.71) | 0.8 (1.48) | 0.5 (0.98) | 1.9 (3.91) | 2.2 (5.66) | 0.8 (1.59)
  Week 12: number analyzed (Participants) | 32 | 28 | 30 | 35 | 36 | 31 | 32
  Week 12 | 1.4 (2.76) | 0.5 (0.96) | 1.3 (2.07) | 1.1 (2.73) | 1.4 (2.65) | 1.3 (2.30) | 1.3 (2.90)
  Week 16: number analyzed (Participants) | 33 | 27 | 30 | 34 | 31 | 31 | 31
  Week 16 | 1.0 (1.72) | 0.6 (1.24) | 0.9 (1.89) | 1.0 (2.19) | 1.5 (2.92) | 1.1 (2.72) | 1.2 (3.32)
  Week 20: number analyzed (Participants) | 27 | 28 | 30 | 34 | 30 | 32 | 32
  Week 20 | 0.8 (1.42) | 0.4 (0.88) | 0.9 (1.75) | 1.6 (3.03) | 1.0 (2.20) | 0.6 (1.54) | 1.1 (2.79)
  Week 24: number analyzed (Participants) | 28 | 28 | 29 | 32 | 28 | 30 | 31
  Week 24 | 0.9 (2.51) | 0.5 (1.17) | 0.8 (1.33) | 1.4 (3.80) | 0.7 (1.74) | 0.9 (1.87) | 1.0 (2.52)
  Week 36: number analyzed (Participants) | 26 | 26 | 31 | 32 | 28 | 31 | 29
  Week 36 | 0.7 (1.46) | 0.7 (1.67) | 1.1 (3.12) | 1.2 (2.30) | 1.4 (3.24) | 1.0 (2.34) | 0.9 (1.45)
  Week 48: number analyzed (Participants) | 26 | 25 | 27 | 31 | 26 | 25 | 24
  Week 48 | 0.6 (1.50) | 0.2 (0.52) | 0.3 (0.72) | 1.0 (2.42) | 0.8 (2.40) | 1.1 (3.24) | 1.1 (2.59)

4. Secondary Outcome: Total Number of New or Newly Enlarging T2-Weighted MRI Lesions
Description: Lesions were measured using T2-weighted proton density MRI scans.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 36, and 48
Population: Randomized participants who had a T2-weighted MRI assessment at the specified time points.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | 4 mg LY2127399 Q4W | 12 mg LY2127399 Q4W | 40 mg LY2127399 Q4W | 120 mg LY2127399 Q4W | 4 mg LY2127399 Q12W | 120 mg LY2127399 Q12W | Placebo
Number analyzed (Participants) | 34 | 33 | 31 | 36 | 36 | 34 | 34
lesions
  Week 4: number analyzed (Participants) | 34 | 31 | 31 | 36 | 35 | 34 | 34
  Week 4 | 1.5 (2.21) | 0.7 (1.39) | 0.7 (1.46) | 0.9 (1.66) | 2.1 (3.48) | 1.4 (2.47) | 2.0 (3.28)
  Week 8: number analyzed (Participants) | 33 | 33 | 31 | 35 | 36 | 32 | 34
  Week 8 | 1.5 (2.60) | 0.9 (2.23) | 1.0 (1.69) | 0.7 (1.13) | 2.4 (4.42) | 2.8 (6.88) | 1.2 (2.21)
  Week 12: number analyzed (Participants) | 32 | 28 | 30 | 35 | 36 | 31 | 32
  Week 12 | 1.7 (3.35) | 1.1 (1.88) | 1.3 (2.01) | 1.3 (2.85) | 2.0 (3.66) | 1.9 (3.45) | 1.7 (3.51)
  Week 16: number analyzed (Participants) | 33 | 27 | 30 | 34 | 31 | 31 | 31
  Week 16 | 1.2 (2.07) | 1.0 (1.85) | 1.4 (2.73) | 1.5 (3.10) | 1.8 (3.49) | 1.7 (4.12) | 1.5 (4.23)
  Week 20: number analyzed (Participants) | 27 | 28 | 30 | 34 | 30 | 32 | 32
  Week 20 | 0.9 (1.66) | 0.8 (1.70) | 1.2 (2.16) | 2.1 (4.40) | 1.6 (4.06) | 1.0 (1.88) | 1.4 (4.20)
  Week 24: number analyzed (Participants) | 28 | 28 | 29 | 32 | 28 | 30 | 31
  Week 24 | 1.0 (2.37) | 0.7 (1.51) | 1.2 (2.42) | 1.7 (4.28) | 1.0 (2.40) | 1.3 (2.79) | 1.5 (3.52)
  Week 36: number analyzed (Participants) | 26 | 26 | 31 | 32 | 28 | 31 | 29
  Week 36 | 1.5 (2.55) | 1.6 (3.02) | 2.4 (4.27) | 2.8 (5.18) | 3.0 (6.64) | 2.8 (4.69) | 1.6 (3.31)
  Week 48: number analyzed (Participants) | 26 | 25 | 28 | 31 | 27 | 25 | 24
  Week 48 | 1.3 (2.56) | 0.4 (0.65) | 1.8 (4.16) | 2.8 (6.04) | 1.7 (3.82) | 1.5 (4.06) | 1.8 (3.84)

5. Secondary Outcome: Total Volume of T2-Weighted MRI Lesions
Description: The total volume of T2-weighted lesions was measured using T2-weighted proton density MRI scans. LS mean was calculated using an ANOVA model.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 36, and 48
Population: Randomized participants who had a T2-weighted MRI assessment at the specified time points.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | 4 mg LY2127399 Q4W | 12 mg LY2127399 Q4W | 40 mg LY2127399 Q4W | 120 mg LY2127399 Q4W | 4 mg LY2127399 Q12W | 120 mg LY2127399 Q12W | Placebo
Number analyzed (Participants) | 34 | 33 | 31 | 36 | 36 | 34 | 34
mL
  Week 4: number analyzed (Participants) | 34 | 31 | 31 | 36 | 35 | 34 | 34
  Week 4 | 8.7 (1.73) | 7.6 (1.81) | 6.3 (1.81) | 8.7 (1.68) | 10.5 (1.71) | 6.8 (1.73) | 7.7 (1.73)
  Week 8: number analyzed (Participants) | 33 | 33 | 31 | 35 | 36 | 32 | 34
  Week 8 | 8.8 (1.74) | 8.0 (1.74) | 6.2 (1.80) | 9.0 (1.69) | 10.1 (1.67) | 7.3 (1.77) | 6.7 (1.72)
  Week 12: number analyzed (Participants) | 32 | 28 | 30 | 35 | 36 | 31 | 32
  Week 12 | 8.8 (1.80) | 7.4 (1.92) | 6.3 (1.86) | 8.9 (1.72) | 10.1 (1.70) | 7.7 (1.83) | 6.7 (1.80)
  Week 16: number analyzed (Participants) | 33 | 27 | 30 | 34 | 31 | 31 | 31
  Week 16 | 8.4 (1.79) | 7.3 (1.97) | 6.3 (1.87) | 8.6 (1.76) | 10.7 (1.84) | 7.6 (1.84) | 6.7 (1.84)
  Week 20: number analyzed (Participants) | 27 | 28 | 30 | 34 | 30 | 32 | 32
  Week 20 | 7.0 (1.89) | 7.7 (1.86) | 6.4 (1.80) | 9.1 (1.69) | 10.4 (1.80) | 7.4 (1.74) | 6.8 (1.74)
  Week 24: number analyzed (Participants) | 28 | 28 | 29 | 32 | 28 | 30 | 31
  Week 24 | 7.3 (1.91) | 7.7 (1.91) | 6.4 (1.88) | 9.7 (1.79) | 10.1 (1.91) | 7.7 (1.85) | 6.9 (1.82)
  Week 36: number analyzed (Participants) | 26 | 26 | 31 | 32 | 28 | 31 | 29
  Week 36 | 7.1 (2.01) | 7.3 (2.01) | 6.8 (1.84) | 9.7 (1.81) | 11.5 (1.94) | 7.2 (1.84) | 6.6 (1.91)
  Week 48: number analyzed (Participants) | 26 | 25 | 28 | 31 | 27 | 25 | 24
  Week 48 | 6.6 (2.01) | 7.7 (2.05) | 7.0 (1.93) | 9.9 (1.84) | 11.5 (1.97) | 6.0 (2.05) | 4.6 (2.09)

6. Secondary Outcome: Expanded Disability Status Scale (EDSS)
Description: The EDSS is a rating scale for quantifying disability in multiple sclerosis (MS) participants. The EDSS has 8 functional systems (pyramidal, cerebellar, brain stem, sensory, bowel and bladder, visual, cerebral, and other) each rated on a scale from 0 (normal) to 5 (severe disability) or 0 (normal) to 6 (severe disability). The EDSS score was computed based on an algorithm of these components, and scores ranged from 0.0 (normal neurological exam) to 10.0 (death due to MS) in increments of 0.5.
Time Frame: Weeks 12, 24, and 48
Population: Randomized participants who had EDSS scores at the specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 4 mg LY2127399 Q4W | 12 mg LY2127399 Q4W | 40 mg LY2127399 Q4W | 120 mg LY2127399 Q4W | 4 mg LY2127399 Q12W | 120 mg LY2127399 Q12W | Placebo
Number analyzed (Participants) | 35 | 32 | 30 | 36 | 36 | 34 | 33
units on a scale
  Week 12 | 2.96 (1.146) | 2.75 (1.397) | 2.65 (1.212) | 2.17 (1.493) | 2.54 (1.490) | 2.54 (1.395) | 2.47 (1.457)
  Week 24: number analyzed (Participants) | 29 | 29 | 30 | 32 | 29 | 30 | 31
  Week 24 | 2.91 (0.992) | 2.78 (1.334) | 2.62 (1.250) | 2.17 (1.429) | 2.64 (1.625) | 2.82 (1.283) | 2.77 (1.419)
  Week 48: number analyzed (Participants) | 27 | 26 | 29 | 31 | 27 | 28 | 25
  Week 48 | 2.96 (1.263) | 2.46 (1.612) | 2.74 (1.066) | 2.18 (1.568) | 2.57 (1.505) | 2.73 (1.357) | 2.60 (1.377)

7. Secondary Outcome: Time to First Relapse
Description: A confirmed relapse was defined as the appearance of 1 or more new neurological symptom(s) attributable to MS or the worsening of 1 or more previously observed symptoms. This change in clinical state was to last at least 48 hours and be immediately preceded by an improving neurological state of at least 30 days from onset of previous relapse. New or worsening neurological symptoms were accompanied by objective EDSS changes on examination (an increase from baseline of at least 1 point on the EDSS, at least 1 point on 2 EDSS functional systems, or at least 2 points on 1 EDSS functional system). A relapse may or may not have required systemic corticosteroid treatment. If a relapse did not occur during the specified time frame, the time to the first confirmed relapse was censored to the date of the participant's last available visit at or prior to Week 24, Week 48, and Week 48 for the respective time frames.
Time Frame: Baseline through Week 24, Baseline through Week 48, and Week 24 through Week 48
Population: Randomized participants who had a relapse assessment for the specified time periods. Twenty-one (21), 24, 24, 28, 23, 26, and 26 participants were censored in the following arms respectively: 4 mg, 12 mg, 40 mg, and 120 mg LY2127399 Q4W, 4 mg and 120 mg LY2127399 Q12W, and placebo.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 4 mg LY2127399 Q4W | 12 mg LY2127399 Q4W | 40 mg LY2127399 Q4W | 120 mg LY2127399 Q4W | 4 mg LY2127399 Q12W | 120 mg LY2127399 Q12W | Placebo
Number analyzed (Participants) | 35 | 34 | 33 | 36 | 36 | 35 | 35
days
  Baseline through Week 24 | 139.54 (48.949) | 141.56 (51.460) | 154.73 (40.117) | 153.72 (32.753) | 140.06 (53.970) | 151.23 (40.717) | 148.37 (49.911)
  Baseline through Week 48 | 243.57 (119.991) | 242.68 (123.805) | 286.85 (99.004) | 279.17 (100.955) | 241.97 (119.871) | 272.23 (105.653) | 276.46 (112.039)
  Week 24 through Week 48: number analyzed (Participants) | 29 | 28 | 30 | 33 | 28 | 30 | 31
  Week 24 through Week 48 | 144.38 (46.900) | 144.46 (49.736) | 154.33 (51.892) | 163.39 (22.685) | 150.32 (36.685) | 148.07 (51.075) | 161.23 (16.346)

8. Secondary Outcome: Percentage of Relapse-Free Participants
Description: A confirmed relapse was defined as the appearance of 1 or more new neurological symptom(s) attributable to MS or the worsening of 1 or more previously observed symptoms. This change in clinical state was to last at least 48 hours and be immediately preceded by an improving neurological state of at least 30 days from onset of previous relapse. New or worsening neurological symptoms were accompanied by objective EDSS changes on examination (an increase from baseline of at least 1 point on the EDSS, at least 1 point on 2 EDSS functional systems, or at least 2 points on 1 EDSS functional system). A relapse may or may not have required systemic corticosteroid treatment. Percentage of relapse-free participants=[(number of participants who did not relapse)/(number of pts assessed)]*100.
Time Frame: Week 24, Week 48, end of study treatment [Week 24 or early discontinuation (ED)], and end of follow-up (Week 48 or ED)
Population: Randomized participants who had a relapse assessment at the specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | 4 mg LY2127399 Q4W | 12 mg LY2127399 Q4W | 40 mg LY2127399 Q4W | 120 mg LY2127399 Q4W | 4 mg LY2127399 Q12W | 120 mg LY2127399 Q12W | Placebo
Number analyzed (Participants) | 35 | 34 | 33 | 36 | 36 | 35 | 35
percentage of participants
  Week 24: number analyzed (Participants) | 29 | 29 | 31 | 33 | 29 | 31 | 31
  Week 24 | 72.4 | 82.8 | 77.4 | 84.8 | 79.3 | 83.9 | 83.9
  Week 48: number analyzed (Participants) | 27 | 26 | 31 | 32 | 28 | 29 | 27
  Week 48 | 70.4 | 73.1 | 64.5 | 75.0 | 67.9 | 72.4 | 77.8
  End of Treatment | 74.3 | 76.5 | 78.8 | 83.3 | 75.0 | 80.0 | 82.9
  End of Follow-Up | 68.6 | 67.6 | 66.7 | 77.8 | 63.9 | 65.7 | 77.1

9. Secondary Outcome: Annualized Relapse Rate (ARR) at Week 24 and Week 48
Description: The number of confirmed relapses per year, ARR=[(number of relapses from baseline through Week 24 or baseline through Week 48)/(the time in days between the same interval)]*365.25. A confirmed relapse was defined as the appearance of 1 or more new neurological symptom(s) attributable to MS or the worsening of 1 or more previously observed symptoms. This change in clinical state was to last at least 48 hours and be immediately preceded by an improving neurological state of at least 30 days from onset of previous relapse. New or worsening neurological symptoms were accompanied by objective EDSS changes on examination (an increase from baseline of at least 1 point on the EDSS, at least 1 point on 2 EDSS functional systems, or at least 2 points on 1 EDSS functional system). A relapse may or may have not required systemic corticosteroid treatment.
Time Frame: Baseline through Week 24 and Baseline through Week 48
Population: Randomized participants who had a relapse assessment for the specified time periods.
Measure: Mean (Standard Deviation); unit: relapses per year
Arm/Group | 4 mg LY2127399 Q4W | 12 mg LY2127399 Q4W | 40 mg LY2127399 Q4W | 120 mg LY2127399 Q4W | 4 mg LY2127399 Q12W | 120 mg LY2127399 Q12W | Placebo
Number analyzed (Participants) | 35 | 34 | 33 | 36 | 36 | 35 | 35
relapses per year
  Week 24 | 0.75 (1.568) | 0.80 (1.830) | 0.33 (0.787) | 0.38 (0.856) | 0.67 (1.536) | 0.51 (1.205) | 0.71 (2.844)
  Week 48 | 0.67 (1.463) | 0.64 (1.284) | 0.36 (0.645) | 0.24 (0.461) | 0.56 (0.966) | 0.53 (0.936) | 0.66 (2.805)

10. Secondary Outcome: Multiple Sclerosis Functional Composite Scale (MSFC)
Description: The MSFC is a composite scale consisting of 3 components [Timed 25-Foot Walk, 9-Hole Peg Test (9-HPT), and 3-Second Paced Auditory Serial Addition Test (PASAT-3)]. The Timed 25-Foot Walk was a quantitative measure of lower extremity function. The 9-HPT was a quantitative measure of upper extremity (arm and hand) function. The PASAT-3 was a measure of cognitive function that specifically assessed auditory information processing speed and flexibility, as well as calculation ability. Component scores ranged from 0 to 60 and were converted to standard scores (z-scores). The MSFC score was calculated as the average of the 3 standardized component scores. Higher MSFC scores reflected better neurological function.
Time Frame: Weeks 12, 24, and 48
Population: Randomized participants who had MSFC scores at the specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 4 mg LY2127399 Q4W | 12 mg LY2127399 Q4W | 40 mg LY2127399 Q4W | 120 mg LY2127399 Q4W | 4 mg LY2127399 Q12W | 120 mg LY2127399 Q12W | Placebo
Number analyzed (Participants) | 35 | 32 | 31 | 35 | 34 | 34 | 32
units on a scale
  Week 12: number analyzed (Participants) | 35 | 32 | 30 | 35 | 34 | 34 | 32
  Week 12 | 0.11 (0.821) | 0.08 (0.511) | -0.02 (0.385) | 0.06 (0.396) | -0.02 (0.471) | 0.26 (0.870) | 0.39 (0.955)
  Week 24: number analyzed (Participants) | 28 | 28 | 31 | 33 | 28 | 31 | 30
  Week 24 | 0.05 (0.741) | 0.11 (0.461) | 0.02 (0.369) | 0.17 (0.547) | -0.06 (0.316) | 0.15 (0.707) | 0.24 (0.606)
  Week 48: number analyzed (Participants) | 27 | 25 | 29 | 31 | 28 | 28 | 25
  Week 48 | -0.11 (0.504) | 0.07 (0.471) | 0.04 (0.350) | 0.08 (0.332) | 0.03 (0.321) | 0.10 (0.388) | 0.13 (0.344)

11. Secondary Outcome: Visual Analog Scale (VAS) of Wellbeing
Description: The VAS is a 100-millimeter (mm) horizontal line marked with 0 mm = "poor" and 100 mm = "excellent." Participants were asked to assess their wellbeing by making a vertical mark on the scale. The score was computed as the distance from 0 mm to the vertical mark.
Time Frame: Weeks 12, 24, and 48
Population: Randomized participants who had VAS of Wellbeing scores at the specified time points.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 4 mg LY2127399 Q4W | 12 mg LY2127399 Q4W | 40 mg LY2127399 Q4W | 120 mg LY2127399 Q4W | 4 mg LY2127399 Q12W | 120 mg LY2127399 Q12W | Placebo
Number analyzed (Participants) | 35 | 32 | 31 | 36 | 36 | 33 | 33
mm
  Week 12: number analyzed (Participants) | 35 | 32 | 30 | 36 | 36 | 33 | 33
  Week 12 | 55.86 (24.686) | 61.09 (20.934) | 63.20 (24.864) | 65.78 (24.114) | 59.67 (21.511) | 64.67 (22.235) | 60.18 (20.430)
  Week 24: number analyzed (Participants) | 28 | 29 | 31 | 33 | 29 | 31 | 30
  Week 24 | 58.86 (22.874) | 54.79 (23.665) | 63.26 (18.630) | 61.42 (23.829) | 57.76 (23.257) | 60.84 (23.602) | 55.70 (26.785)
  Week 48: number analyzed (Participants) | 26 | 26 | 29 | 31 | 28 | 28 | 25
  Week 48 | 59.77 (26.288) | 56.19 (26.872) | 62.93 (25.201) | 65.29 (24.487) | 52.71 (23.434) | 56.39 (26.720) | 64.48 (24.985)

12. Secondary Outcome: 16-Item Quick Inventory for Depressive Symptomatology Self Report (QIDS-SR16)
Description: The QIDS-SR16 is a 16-item participant-rated measure of depressive symptomatology. Each item corresponds to 1 of 9 criterion domains for depression: change in sleep disturbance [question (Q) 1 through Q4], sad mood (Q5), decrease or increase in appetite and weight (Q6 through Q9), concentration (Q10), self-criticism (Q11), suicidal ideation (Q12), interest (Q13), energy/fatigue (Q14), and psychomotor agitation and retardation (Q15 and Q16). Each question was scored 0 (no problems) to 3 (increased symptoms). The total score=(the highest score from Q1 through Q4)+(Q5 score)+(the highest score from Q6 through Q9)+(the total score for each Q10 through Q14)+(the highest score from Q15 and Q16). A total score of 0 through 5 was considered no depression likely, 6 through 10 was mild depression, 11 through 15 was moderate depression, 16 through 20 was severe depression, and 21 or over was very severe depression.
Time Frame: Weeks 12, 24, and 48
Population: Randomized participants who had QIDS-SR16 scores at the specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 4 mg LY2127399 Q4W | 12 mg LY2127399 Q4W | 40 mg LY2127399 Q4W | 120 mg LY2127399 Q4W | 4 mg LY2127399 Q12W | 120 mg LY2127399 Q12W | Placebo
Number analyzed (Participants) | 34 | 32 | 31 | 36 | 36 | 33 | 32
units on a scale
  Week 12: number analyzed (Participants) | 34 | 32 | 30 | 36 | 36 | 33 | 32
  Week 12 | 7.79 (4.766) | 6.78 (4.668) | 7.13 (5.322) | 5.94 (3.695) | 7.47 (3.676) | 6.42 (4.000) | 7.38 (4.577)
  Week 24: number analyzed (Participants) | 28 | 28 | 31 | 33 | 29 | 31 | 30
  Week 24 | 7.25 (5.082) | 6.43 (4.717) | 6.52 (3.906) | 6.30 (4.660) | 7.21 (3.867) | 6.84 (3.934) | 6.23 (3.441)
  Week 48: number analyzed (Participants) | 26 | 26 | 28 | 31 | 28 | 28 | 25
  Week 48 | 6.38 (4.491) | 5.54 (3.723) | 6.82 (5.143) | 5.74 (3.651) | 7.68 (5.004) | 7.43 (4.272) | 6.20 (4.537)

13. Secondary Outcome: Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) Component Scores
Description: The SF-36 was a 36-item, health-related survey that assessed participant's quality of life on 8 domains: physical functioning, bodily pain, role limitations due to physical problems, role limitations due to emotional problems, general health, mental health, social functioning, vitality and 2 component scores (mental and physical health). Domain scores were calculated by summing individual items for each domain and transforming scores into 0 to 100 scale; higher scores indicated better health status or function. The mental component summary (MCS) score, based on SF-36 domains, consisted of social functioning, vitality, mental health, and role-emotional scales (range: 0 to 100). The physical component summary (PCS) score, based on SF-36 domains, consisted of physical functioning, bodily pain, role-physical, and general health scales (range: 0 to 100).
Time Frame: Weeks 12, 24, and 48
Population: Randomized participants who had SF-36 component scores at the specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 4 mg LY2127399 Q4W | 12 mg LY2127399 Q4W | 40 mg LY2127399 Q4W | 120 mg LY2127399 Q4W | 4 mg LY2127399 Q12W | 120 mg LY2127399 Q12W | Placebo
Number analyzed (Participants) | 35 | 32 | 31 | 36 | 36 | 33 | 33
units on a scale
  PCS, Week 12: number analyzed (Participants) | 35 | 32 | 30 | 36 | 36 | 33 | 33
  PCS, Week 12 | 40.96 (10.673) | 45.53 (9.511) | 44.30 (10.298) | 45.57 (10.716) | 42.80 (9.638) | 42.29 (9.962) | 43.12 (11.656)
  MCS, Week 12: number analyzed (Participants) | 35 | 32 | 30 | 36 | 36 | 33 | 33
  MCS, Week 12 | 42.86 (11.410) | 43.94 (10.736) | 44.62 (13.547) | 48.62 (11.023) | 44.10 (11.675) | 49.08 (9.108) | 46.93 (9.889)
  PCS, Week 24: number analyzed (Participants) | 29 | 29 | 31 | 33 | 29 | 30 | 30
  PCS, Week 24 | 44.08 (9.421) | 44.22 (8.118) | 41.66 (9.927) | 46.30 (9.862) | 44.10 (9.766) | 43.11 (9.890) | 43.81 (10.568)
  MCS, Week 24: number analyzed (Participants) | 29 | 29 | 31 | 33 | 29 | 30 | 30
  MCS, Week 24 | 44.20 (11.836) | 46.95 (10.270) | 46.20 (10.405) | 47.48 (13.101) | 44.90 (11.217) | 46.52 (10.661) | 46.29 (10.150)
  PCS, Week 48: number analyzed (Participants) | 26 | 26 | 29 | 31 | 27 | 28 | 24
  PCS, Week 48 | 44.17 (10.496) | 43.21 (9.144) | 42.43 (9.400) | 47.72 (9.593) | 42.59 (9.011) | 41.22 (12.093) | 44.78 (10.020)
  MCS, Week 48: number analyzed (Participants) | 26 | 26 | 29 | 31 | 27 | 28 | 24
  MCS, Week 48 | 46.40 (11.290) | 49.69 (9.131) | 45.66 (12.016) | 47.89 (13.543) | 44.75 (11.838) | 46.03 (10.618) | 46.85 (10.793)

14. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration-Time Curve for Dosing Interval at Steady State (AUCtau,ss)
Description: AUCtau,ss was obtained by conducting a simulation consisting of 1000 participants, which were then used to determine the noncompartmental PK parameters for each regimen.
Time Frame: Week 0: Day 1, 2, or 3 and Weeks 1, 4, 8, 12, 16, 20, 24, 30, 36, and 40.
Population: Randomized participants who had evaluable PK data.
Measure: Median (Standard Deviation); unit: micrograms/milliliter*hours (mcg/mL*h)
Arm/Group | 4 mg LY2127399 Q4W | 12 mg LY2127399 Q4W | 40 mg LY2127399 Q4W | 120 mg LY2127399 Q4W | 4 mg LY2127399 Q12W | 120 mg LY2127399 Q12W
Number analyzed (Participants) | 35 | 34 | 33 | 36 | 36 | 35
micrograms/milliliter*hours (mcg/mL*h) | 161 (127) | 724 (569) | 4405 (2010) | 16603 (5444) | 146 (108) | 13608 (5746)

15. Secondary Outcome: Percentage of Participants With Anti-LY2127399 Antibodies [Anti-Drug Antibodies (ADA)]
Description: The percentage of participants with ADA=[(number of participants who had ADA)/(number of participants assessed)]*100.
Time Frame: Baseline, Weeks 4, 12, 24, 48, 60, 72, 84, 96, and 108
Population: Randomized participants who had an ADA assessment at the specified time periods.
Measure: Number; unit: percentage of participants
Arm/Group | 4 mg LY2127399 Q4W | 12 mg LY2127399 Q4W | 40 mg LY2127399 Q4W | 120 mg LY2127399 Q4W | 4 mg LY2127399 Q12W | 120 mg LY2127399 Q12W | Placebo
Number analyzed (Participants) | 35 | 33 | 33 | 34 | 36 | 35 | 35
percentage of participants
  Baseline, Positive ADA: number analyzed (Participants) | 35 | 33 | 33 | 34 | 35 | 34 | 33
  Baseline, Positive ADA | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4, Positive ADA | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12, Positive ADA: number analyzed (Participants) | 34 | 32 | 30 | 33 | 34 | 31 | 33
  Week 12, Positive ADA | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 24, Positive ADA: number analyzed (Participants) | 29 | 29 | 30 | 33 | 29 | 30 | 31
  Week 24, Positive ADA | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 48, Positive ADA: number analyzed (Participants) | 26 | 26 | 29 | 31 | 26 | 27 | 25
  Week 48, Positive ADA | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 60, Positive ADA: number analyzed (Participants) | 18 | 24 | 22 | 26 | 26 | 23 | 20
  Week 60, Positive ADA | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 72, Positive ADA: number analyzed (Participants) | 16 | 23 | 23 | 26 | 24 | 21 | 17
  Week 72, Positive ADA | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 84, Positive ADA: number analyzed (Participants) | 3 | 7 | 7 | 12 | 4 | 7 | 2
  Week 84, Positive ADA | 0 | 0 | 0 | 0 | 25.0 | 0 | 0
  Week 96, Positive ADA: number analyzed (Participants) | 0 | 7 | 6 | 12 | 3 | 7 | 2
  Week 96, Positive ADA |  | 0 | 0 | 0 | 0 | 0 | 0
  Week 108, Positive ADA: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Week 108, Positive ADA |  |  |  | 0 |  |  |

16. Secondary Outcome: Pharmacodynamics: Change From Baseline in Peripheral Blood B Cell Subsets (Absolute Cell Counts)
Description: Cell surface marker cluster designation (CD)19, CD27, and immunoglobulin D (IgD) expression levels were used to define the various B cell subsets. Cell surface markers were defined as being either present (+) or absent (-). Peripheral blood B cell subsets included: mature naive B cells (CD19+IgD+CD27-); immature/transitional (immature/tran) B cells (CD19+IgD-CD27-); switched memory B cells (CD19+IgD-CD27+); and non-switched memory B cells (CD19+IgD+CD27+). A positive or negative change indicated an increase or decrease, respectively in B cell count.
Time Frame: Baseline, Day 2, Weeks (Wks) 1, 4, 12, 24, 36, and 48
Population: Randomized participants who had peripheral blood B cell subset cell counts at the specified time points.
Measure: Mean (Standard Deviation); unit: cells per microliter (cells/µL)
Arm/Group | 4 mg LY2127399 Q4W | 12 mg LY2127399 Q4W | 40 mg LY2127399 Q4W | 120 mg LY2127399 Q4W | 4 mg LY2127399 Q12W | 120 mg LY2127399 Q12W | Placebo
Number analyzed (Participants) | 28 | 29 | 29 | 32 | 32 | 30 | 30
cells per microliter (cells/µL)
  Mature Naive, Day 2: number analyzed (Participants) | 28 | 23 | 28 | 30 | 30 | 27 | 29
  Mature Naive, Day 2 | 18.2 (51.9) | 23.8 (35.7) | 26.9 (89.3) | 28.3 (93.4) | 18.6 (49.3) | 16.3 (69.7) | -23.5 (68.3)
  Mature Naive, Wk 1: number analyzed (Participants) | 28 | 29 | 28 | 30 | 32 | 26 | 28
  Mature Naive, Wk 1 | 13.7 (71.3) | 30.2 (69.5) | 27.8 (64.3) | 13.8 (83.0) | 38.5 (51.1) | 30.2 (74.1) | -0.9 (49.2)
  Mature Naive, Wk 4: number analyzed (Participants) | 25 | 29 | 29 | 32 | 27 | 30 | 26
  Mature Naive, Wk 4 | -24.7 (84.7) | -48.0 (49.5) | -54.8 (62.0) | -54.9 (80.1) | -18.9 (30.9) | -73.5 (69.7) | -10.4 (69.7)
  Mature Naive, Wk 12: number analyzed (Participants) | 27 | 27 | 26 | 28 | 29 | 30 | 30
  Mature Naive, Wk 12 | -55.9 (68.7) | -77.0 (57.0) | -116.9 (115.0) | -108.5 (97.4) | -4.2 (42.3) | -130.4 (105.4) | 5.2 (82.8)
  Mature Naive, Wk 24: number analyzed (Participants) | 23 | 24 | 25 | 26 | 23 | 23 | 24
  Mature Naive, Wk 24 | -83.0 (93.3) | -92.7 (72.8) | -143.9 (127.2) | -122.9 (102.3) | -9.0 (62.9) | -149.9 (125.5) | 10.0 (124.5)
  Mature Naive, Wk 36: number analyzed (Participants) | 22 | 23 | 26 | 29 | 26 | 28 | 25
  Mature Naive, Wk 36 | -40.4 (106.1) | -78.9 (78.9) | -147.0 (134.9) | -130.7 (102.3) | -3.0 (66.7) | -118.3 (131.8) | 9.7 (99.9)
  Mature Naive, Wk 48: number analyzed (Participants) | 20 | 20 | 24 | 26 | 24 | 24 | 22
  Mature Naive, Wk 48 | -7.0 (119.3) | -65.7 (101.4) | -118.0 (136.6) | -130.6 (110.5) | 1.5 (69.9) | -92.7 (133.0) | -5.5 (59.9)
  Immature/Tran, Day 2: number analyzed (Participants) | 28 | 23 | 28 | 30 | 30 | 27 | 29
  Immature/Tran, Day 2 | 2.3 (5.4) | 2.0 (6.0) | 0.5 (3.7) | 0.1 (6.8) | 1.4 (4.5) | -4.9 (25.9) | 0.1 (3.5)
  Immature/Tran, Wk 1: number analyzed (Participants) | 28 | 29 | 28 | 30 | 32 | 26 | 28
  Immature/Tran, Wk 1 | 3.7 (10.5) | 1.8 (7.1) | 3.4 (8.5) | 1.9 (9.5) | 3.2 (5.3) | -3.8 (27.6) | -0.3 (4.7)
  Immature/Tran, Wk 4: number analyzed (Participants) | 25 | 29 | 29 | 32 | 27 | 30 | 26
  Immature/Tran, Wk 4 | 1.0 (5.5) | 0.9 (7.0) | 3.8 (13.2) | -0.6 (4.4) | 0.2 (4.0) | -4.8 (25.1) | 3.3 (13.3)
  Immature/Tran Wk 12: number analyzed (Participants) | 27 | 27 | 26 | 28 | 29 | 30 | 30
  Immature/Tran Wk 12 | -0.4 (5.2) | 0.2 (8.3) | -1.0 (4.4) | -2.0 (6.1) | -0.2 (4.3) | -6.4 (26.0) | 2.0 (7.6)
  Immature/Tran Wk 24: number analyzed (Participants) | 23 | 24 | 25 | 26 | 23 | 23 | 24
  Immature/Tran Wk 24 | 2.0 (6.4) | -0.3 (9.0) | -1.7 (4.3) | -2.8 (6.9) | 1.4 (10.8) | -8.3 (29.5) | 0.4 (4.3)
  Immature/Tran, Wk 36: number analyzed (Participants) | 22 | 23 | 26 | 29 | 26 | 28 | 25
  Immature/Tran, Wk 36 | 1.5 (8.7) | 0.1 (6.2) | -3.7 (3.8) | -2.9 (7.7) | 1.8 (7.5) | -9.2 (26.4) | 1.4 (3.6)
  Immature/Tran, Wk 48: number analyzed (Participants) | 20 | 20 | 24 | 26 | 24 | 24 | 22
  Immature/Tran, Wk 48 | 2.9 (8.8) | 1.8 (8.9) | -2.0 (5.1) | -4.0 (9.5) | 9.1 (21.8) | -10.3 (28.0) | 1.3 (6.1)
  Switched Memory, Day 2: number analyzed (Participants) | 28 | 23 | 28 | 30 | 30 | 27 | 29
  Switched Memory, Day 2 | 14.2 (19.3) | 8.0 (19.7) | 8.1 (11.8) | 0.5 (30.5) | 5.5 (12.9) | 7.9 (17.2) | 0.1 (15.0)
  Switched Memory, Wk 1: number analyzed (Participants) | 28 | 29 | 28 | 30 | 32 | 26 | 28
  Switched Memory, Wk 1 | 27.1 (25.9) | 26.0 (24.8) | 26.9 (27.7) | 15.0 (31.0) | 21.8 (18.9) | 28.2 (30.5) | 2.0 (19.2)
  Switched Memory, Wk 4: number analyzed (Participants) | 25 | 29 | 29 | 32 | 27 | 30 | 26
  Switched Memory, Wk 4 | 12.5 (31.6) | 20.5 (19.7) | 28.6 (26.3) | 18.9 (30.7) | -0.1 (18.1) | 31.9 (30.0) | 0.7 (20.3)
  Switched Memory, Wk 12: number analyzed (Participants) | 27 | 27 | 26 | 28 | 29 | 30 | 30
  Switched Memory, Wk 12 | 7.0 (16.4) | 23.5 (20.9) | 26.2 (22.8) | 22.1 (22.3) | -1.9 (16.0) | 15.8 (30.0) | 5.4 (28.3)
  Switched Memory, Wk 24: number analyzed (Participants) | 23 | 24 | 25 | 26 | 23 | 23 | 24
  Switched Memory, Wk 24 | 12.3 (32.8) | 24.5 (26.4) | 23.8 (23.4) | 16.8 (31.0) | 8.9 (22.8) | 17.4 (31.3) | 3.0 (25.3)
  Switched Memory, Wk 36: number analyzed (Participants) | 22 | 23 | 26 | 29 | 26 | 28 | 25
  Switched Memory, Wk 36 | 8.9 (63.2) | -10.3 (21.1) | -9.1 (15.6) | 6.5 (41.0) | -1.0 (24.5) | -18.7 (26.4) | 1.5 (16.6)
  Switched Memory, Wk 48: number analyzed (Participants) | 20 | 20 | 24 | 26 | 24 | 24 | 22
  Switched Memory, Wk 48 | 15.0 (45.9) | -7.3 (33.6) | -13.0 (18.3) | -20.4 (38.7) | 11.0 (40.0) | -16.9 (36.2) | -4.1 (25.1)
  Non-Switched Memory, Day 2: number analyzed (Participants) | 28 | 23 | 28 | 30 | 30 | 27 | 29
  Non-Switched Memory, Day 2 | 7.7 (13.4) | 3.8 (10.7) | 11.4 (17.8) | 9.0 (14.2) | 6.7 (19.5) | 7.8 (18.0) | 0.6 (10.8)
  Non-Switched Memory, Wk 1: number analyzed (Participants) | 28 | 29 | 28 | 30 | 32 | 26 | 28
  Non-Switched Memory, Wk 1 | 12.3 (15.9) | 20.3 (30.4) | 19.4 (14.9) | 16.6 (14.9) | 15.4 (18.6) | 18.3 (15.9) | 4.1 (13.2)
  Non-Switched Memory, Wk 4: number analyzed (Participants) | 25 | 29 | 29 | 32 | 27 | 30 | 26
  Non-Switched Memory, Wk 4 | 3.2 (17.6) | 13.8 (16.8) | 16.6 (17.2) | 22.3 (27.1) | 1.8 (8.4) | 17.3 (16.5) | -1.3 (10.7)
  Non-Switched Memory Wk 12: number analyzed (Participants) | 27 | 27 | 26 | 28 | 29 | 30 | 30
  Non-Switched Memory Wk 12 | 4.9 (15.2) | 24.2 (49.7) | 18.7 (21.9) | 14.8 (15.2) | -0.6 (11.8) | 8.6 (21.5) | -0.4 (12.0)
  Non-Switched Memory Wk 24 (n=23,24,25,26,23,23,24): number analyzed (Participants) | 23 | 24 | 25 | 26 | 23 | 23 | 24
  Non-Switched Memory Wk 24 (n=23,24,25,26,23,23,24) | 2.2 (19.7) | 15.6 (34.5) | 17.3 (24.5) | 15.3 (17.4) | 3.0 (20.4) | 10.4 (35.6) | 2.5 (14.8)
  Non-Switched Memory, Wk 36: number analyzed (Participants) | 22 | 23 | 26 | 29 | 26 | 28 | 25
  Non-Switched Memory, Wk 36 | 1.5 (38.0) | -9.0 (24.6) | -8.5 (11.0) | 9.6 (36.5) | -1.2 (18.2) | -15.1 (28.7) | -1.0 (13.4)
  Non-Switched Memory, Wk 48: number analyzed (Participants) | 20 | 20 | 24 | 26 | 24 | 24 | 22
  Non-Switched Memory, Wk 48 | 22.9 (88.4) | -4.4 (32.3) | -13.3 (9.3) | -7.4 (38.5) | -3.0 (17.7) | -17.3 (19.9) | -5.8 (16.7)

ADVERSE EVENTS:
Time Frame: Baseline through end of study treatment (up to and through Week 24 or ED) and post-study treatment follow-up (start of Week 25 or ED) through study completion (up to and through Week 48) plus long-term follow-up (up to and through Week 108)
Description: Randomized participants who received any amount of study drug.
Groups:
- 4 mg LY2127399 Q4W, Treatment: Adverse Events (AEs) reported during study treatment (up to Week 24).
  LY2127399: 4 mg subcutaneous injection Q4W for 24 weeks (Weeks 0, 4, 8, 12, 16, and 20).
- 12 mg LY2127399 Q4W, Treatment: AEs reported during study treatment (up to Week 24).
  LY2127399: 12 mg subcutaneous injection Q4W for 24 weeks.
- 40 mg LY2127399 Q4W, Treatment: AEs reported during study treatment (up to Week 24).
  LY2127399: 40 mg subcutaneous injection Q4W for 24 weeks.
- 120 mg LY2127399 Q4W, Treatment: AEs reported during study treatment (up to Week 24).
  LY2127399: 120 mg subcutaneous injection Q4W for 24 weeks.
- 4 mg LY2127399 Q12W, Treatment: AEs reported during study treatment (up to Week 24).
  LY2127399: 4 mg subcutaneous injection Q12W for 24 weeks (Weeks 0 and 12).
  Placebo: Subcutaneous injection Q4W for 24 weeks (except Weeks 0 and 12).
- 120 mg LY2127399 Q12W, Treatment: AEs reported during study treatment (up to Week 24).
  LY2127399: 120 mg subcutaneous injection Q12W for 24 weeks (Weeks 0 and 12).
  Placebo: Subcutaneous injection every Q4W for 24 weeks (except Weeks 0 and 12).
- Placebo, Treatment: AEs reported during study treatment (up to Week 24).
  Placebo: Subcutaneous injection Q4W for 24 weeks.
- 4 mg LY2127399 Q4W, Post-Study Treatment Follow-Up: AEs that started or worsened after Week 24 or ED through long-term follow-up (up to Week 108) for participants who received a 4 mg LY2127399 subcutaneous injection Q4W for 24 weeks.
  No study drug was administered during the post-study treatment follow-up.
- 12 mg LY2127399 Q4W, Post-Study Treatment Follow-Up: AEs that started or worsened after Week 24 or ED through long-term follow-up (up to Week 108) for participants who received a 12 mg LY2127399 subcutaneous injection Q4W for 24 weeks.
  No study drug was administered during the post-study treatment follow-up.
- 40 mg LY2127399 Q4W, Post-Study Treatment Follow-Up: AEs that started or worsened after Week 24 or ED through long-term follow-up (up to Week 108) for participants who received a 40 mg LY2127399 subcutaneous injection Q4W for 24 weeks.
  No study drug was administered during the post-study treatment follow-up.
- 120 mg LY2127399 Q4W, Post-Study Treatment Follow-Up: AEs that started or worsened after Week 24 or ED through long-term follow-up (up to Week 108) for participants who received a 120 mg LY2127399 subcutaneous injection Q4W for 24 weeks.
  No study drug was administered during the post-study treatment follow-up.
- 4 mg LY2127399 Q12W, Post-Study Treatment Follow-Up: AEs that started or worsened after Week 24 or ED through long-term follow-up (up to Week 108) for participants who received a 4 mg LY2127399 subcutaneous injection Q12W for 24 weeks (Weeks 0 and 12) and a placebo subcutaneous injection Q4W for 24 weeks (except Weeks 0 and 12).
  No study drug was administered during the post-study treatment follow-up.
- 120 mg LY2127399 Q12W, Post-Study Treatment Follow-Up: AEs that started or worsened after Week 24 or ED through long-term follow-up (up to Week 108) for participants who received a120 mg LY2127399 subcutaneous injection Q12W for 24 weeks (Weeks 0 and 12) and a placebo subcutaneous injection Q4W for 24 weeks (except Weeks 0 and 12).
  No study drug was administered during the post-study treatment follow-up.
- Placebo, Post-Study Treatment Follow-Up: AEs that started or worsened after Week 24 or ED through long-term follow-up (up to Week 108) for participants who received a placebo subcutaneous injection Q4W for 24 weeks.
  No study drug was administered during the post-study treatment follow-up.
Arm/Group | 4 mg LY2127399 Q4W, Treatment | 12 mg LY2127399 Q4W, Treatment | 40 mg LY2127399 Q4W, Treatment | 120 mg LY2127399 Q4W, Treatment | 4 mg LY2127399 Q12W, Treatment | 120 mg LY2127399 Q12W, Treatment | Placebo, Treatment | 4 mg LY2127399 Q4W, Post-Study Treatment Follow-Up | 12 mg LY2127399 Q4W, Post-Study Treatment Follow-Up | 40 mg LY2127399 Q4W, Post-Study Treatment Follow-Up | 120 mg LY2127399 Q4W, Post-Study Treatment Follow-Up | 4 mg LY2127399 Q12W, Post-Study Treatment Follow-Up | 120 mg LY2127399 Q12W, Post-Study Treatment Follow-Up | Placebo, Post-Study Treatment Follow-Up
Serious Adverse Events (participants affected / at risk) | 2/35 | 4/34 | 2/34 | 3/36 | 3/36 | 2/35 | 1/35 | 2/35 | 2/34 | 4/34 | 1/36 | 3/36 | 5/35 | 2/35
Other Adverse Events (participants affected / at risk) | 21/35 | 22/34 | 25/34 | 19/36 | 28/36 | 25/35 | 17/35 | 17/35 | 12/34 | 16/34 | 10/36 | 15/36 | 14/35 | 12/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4 mg LY2127399 Q4W, Treatment (N=35) | 12 mg LY2127399 Q4W, Treatment (N=34) | 40 mg LY2127399 Q4W, Treatment (N=34) | 120 mg LY2127399 Q4W, Treatment (N=36) | 4 mg LY2127399 Q12W, Treatment (N=36) | 120 mg LY2127399 Q12W, Treatment (N=35) | Placebo, Treatment (N=35) | 4 mg LY2127399 Q4W, Post-Study Treatment Follow-Up (N=35) | 12 mg LY2127399 Q4W, Post-Study Treatment Follow-Up (N=34) | 40 mg LY2127399 Q4W, Post-Study Treatment Follow-Up (N=34) | 120 mg LY2127399 Q4W, Post-Study Treatment Follow-Up (N=36) | 4 mg LY2127399 Q12W, Post-Study Treatment Follow-Up (N=36) | 120 mg LY2127399 Q12W, Post-Study Treatment Follow-Up (N=35) | Placebo, Post-Study Treatment Follow-Up (N=35)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEART DISEASE CONGENITAL (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BREAST CANCER IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AXONAL NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BALANCE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MULTIPLE SCLEROSIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 1 (1) | 3 (4) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
PARESIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE PSYCHOSIS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SCHIZOPHRENIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 4 mg LY2127399 Q4W, Treatment (N=35) | 12 mg LY2127399 Q4W, Treatment (N=34) | 40 mg LY2127399 Q4W, Treatment (N=34) | 120 mg LY2127399 Q4W, Treatment (N=36) | 4 mg LY2127399 Q12W, Treatment (N=36) | 120 mg LY2127399 Q12W, Treatment (N=35) | Placebo, Treatment (N=35) | 4 mg LY2127399 Q4W, Post-Study Treatment Follow-Up (N=35) | 12 mg LY2127399 Q4W, Post-Study Treatment Follow-Up (N=34) | 40 mg LY2127399 Q4W, Post-Study Treatment Follow-Up (N=34) | 120 mg LY2127399 Q4W, Post-Study Treatment Follow-Up (N=36) | 4 mg LY2127399 Q12W, Post-Study Treatment Follow-Up (N=36) | 120 mg LY2127399 Q12W, Post-Study Treatment Follow-Up (N=35) | Placebo, Post-Study Treatment Follow-Up (N=35)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LEFT VENTRICULAR HYPERTROPHY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EUSTACHIAN TUBE DYSFUNCTION (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EUSTACHIAN TUBE OBSTRUCTION (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOACUSIS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GOITRE (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIPLOPIA (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRY EYE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE ALLERGY (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE MOVEMENT DISORDER (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE PAIN (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OPTIC NERVE DISORDER (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHOTOPHOBIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UVEITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VISUAL ACUITY REDUCED (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISUAL IMPAIRMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIVERTICULUM (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FAECAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL MOTILITY DISORDER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 4 (6) | 1 (1) | 3 (5) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA ORAL (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHILLS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CYST (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENERGY INCREASED (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FACIAL PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 4 (4) | 4 (4) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
FEELING COLD (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEELING HOT (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAIT DISTURBANCE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERPYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE ERYTHEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE HAEMATOMA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE PAIN (General disorders) | 1 (2) | 4 (8) | 3 (8) | 4 (8) | 1 (2) | 2 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE REACTION (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IRRITABILITY (General disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SENSATION OF FOREIGN BODY (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TEMPERATURE INTOLERANCE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONTRAST MEDIA ALLERGY (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
BRONCHITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CERVICITIS (Infections and infestations) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 1/21 (1) | 0/27 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 0/21 (0) | 0/27 (0) | 0/24 (0) | 0/24 (0)
CYSTITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DERMATITIS INFECTED (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FUNGAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FURUNCLE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEPATITIS B (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES SIMPLEX (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
LARYNGITIS (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTITIS EXTERNA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARONYCHIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINOTRACHEITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (1) | 5 (5) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 4 (5) | 2 (2) | 2 (3) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VAGINAL INFECTION (Infections and infestations) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 1/21 (1) | 0/27 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/22 (0) | 1/27 (1) | 0/21 (0) | 1/27 (1) | 0/24 (0) | 0/24 (0)
VAGINITIS BACTERIAL (Infections and infestations) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 1/21 (1) | 1/27 (2) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/22 (0) | 1/27 (1) | 0/21 (0) | 0/27 (0) | 0/24 (0) | 0/24 (0)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
VIRAL RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
ALLERGIC TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHROPOD STING (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
EXCORIATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (5) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOREIGN BODY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MENISCUS LESION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (6) | 0 (0) | 0 (0) | 2 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AMYLASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CHOLESTEROL INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BODY TEMPERATURE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM QT INTERVAL ABNORMAL (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMOGLOBIN A PRESENT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATITIS B CORE ANTIBODY POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEPATITIS B SURFACE ANTIBODY POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LIPASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINE LEUKOCYTE ESTERASE POSITIVE (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FLUID RETENTION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OBESITY (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE TWITCHING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SENSATION OF HEAVINESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BENIGN UTERINE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 1/21 (1) | 0/27 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 0/21 (0) | 0/27 (0) | 0/24 (0) | 0/24 (0)
APHASIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AREFLEXIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATAXIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BALANCE DISORDER (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
BURNING SENSATION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COGNITIVE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
DROOLING (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSKINESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FACIAL SPASM (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEAD DISCOMFORT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 5 (12) | 3 (5) | 4 (5) | 3 (4) | 2 (2) | 5 (6) | 3 (9) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 1 (3) | 0 (0) | 2 (4) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
MONOPARESIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEURALGIA (Nervous system disorders) | 2 (2) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NYSTAGMUS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OPTIC NEURITIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RADICULOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESTLESS LEGS SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
SENSORY DISTURBANCE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SENSORY LOSS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TENSION HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AFFECT LABILITY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALCOHOL ABUSE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
CLAUSTROPHOBIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 3 (5) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
HALLUCINATION, VISUAL (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NERVOUSNESS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PANIC ATTACK (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SLEEP DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLADDER IRRITATION (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MICTURITION URGENCY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROGENIC BLADDER (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URETHRAL POLYP (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINE FLOW DECREASED (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATROPHIC VULVOVAGINITIS (Reproductive system and breast disorders) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 0/21 (0) | 0/27 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 0/21 (0) | 0/27 (0) | 1/24 (1) | 0/24 (0)
CYSTOCELE (Reproductive system and breast disorders) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 0/21 (0) | 0/27 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 0/21 (0) | 0/27 (0) | 0/24 (0) | 0/24 (0)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 0/21 (0) | 0/27 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 1/21 (2) | 0/27 (0) | 0/24 (0) | 0/24 (0)
EPIDIDYMITIS (Reproductive system and breast disorders) | 0/11 (0) | 0/12 (0) | 0/7 (0) | 1/15 (1) | 0/9 (0) | 0/11 (0) | 0/11 (0) | 0/11 (0) | 0/12 (0) | 0/7 (0) | 0/15 (0) | 0/9 (0) | 0/11 (0) | 0/11 (0)
MENORRHAGIA (Reproductive system and breast disorders) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 0/21 (0) | 1/27 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/22 (0) | 1/27 (1) | 0/21 (0) | 0/27 (0) | 0/24 (0) | 0/24 (0)
MENSTRUATION DELAYED (Reproductive system and breast disorders) | 0/24 (0) | 0/22 (0) | 1/27 (1) | 0/21 (0) | 0/27 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 0/21 (0) | 0/27 (0) | 0/24 (0) | 0/24 (0)
MENSTRUATION IRREGULAR (Reproductive system and breast disorders) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 0/21 (0) | 0/27 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 0/21 (0) | 1/27 (1) | 0/24 (0) | 0/24 (0)
OVARIAN ADHESION (Reproductive system and breast disorders) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 0/21 (0) | 0/27 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 1/21 (1) | 0/27 (0) | 0/24 (0) | 0/24 (0)
OVARIAN CYST (Reproductive system and breast disorders) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 0/21 (0) | 1/27 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/22 (0) | 1/27 (1) | 0/21 (0) | 0/27 (0) | 0/24 (0) | 0/24 (0)
VULVOVAGINAL DISCOMFORT (Reproductive system and breast disorders) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 1/21 (1) | 0/27 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/22 (0) | 0/27 (0) | 0/21 (0) | 0/27 (0) | 0/24 (0) | 0/24 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 (9) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATION ABNORMAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROAT TIGHTNESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAIR TEXTURE ABNORMAL (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LICHEN PLANUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SCAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN SWELLING (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLUSHING (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL COLDNESS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHLEBITIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VENOUS INSUFFICIENCY (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VENOUS STENOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days